CLINICAL TRIAL: NCT05657964
Title: A Randomized Comparative Effectiveness Trial of Two Postural Therapies for People With Chronic Lower Back Pain (cLBP)-Gokhale Project
Brief Title: Randomized Trial for cLBP (Gokhale Project)
Acronym: Gokhale
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matthew W Smuck, Assoc Professor, Stanford University
Other Study IDs: 60640
Record Dates: First submitted 2022-11-30; First posted 2022-12-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lower Back Pain Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gokhale ARM: Participants enrolled in the Gokhale Arm will be provided the Gokhale PostureTracker, a wearable posture monitoring sensor developed for interactive posture coaching, and a loaner smartphone with pre-installed App. Participants will be provided instruction to apply the sensor on their lumbar area and receive real-time visual feedback on their posture kinematic during the class. Participants can also perform normal daily activities while wearing the device. Data collected by the sensor will be sent to a HIPAA compliance server and shared with Stanford researchers.
  Interventions: Device: Gokhale sensor
- Physical Therapy ARM: Participants randomized into the standard care/physical therapy (PT) arm will similarly receive a standardized PT prescription during a 6-12 weeks period, meeting 1-2 times per week, to include posture education and training, therapeutic exercise instructions and development of an independent home exercise program.

INTERVENTIONS:
Device: Gokhale sensor — Participants enrolled in the Gokhale Arm will be provided the Gokhale PostureTracker, a wearable posture monitoring sensor developed for interactive posture coaching, and a loaner smartphone with pre-installed App. Participants will be provided instruction to apply the sensor on their lumbar area and receive real-time visual feedback on their posture kinematic during the class. Participants can also perform normal daily activities while wearing the device. Data collected by the sensor will be sent to a HIPAA compliance server and shared with Stanford researchers.
  Other Names: Only for Gokhale ARM
  Groups: Gokhale ARM

SUMMARY:
The study aims to compare the effectiveness of the Gokhale Method posture therapy for low back pain (LBP) management to standard physical therapy (PT) with posture training. The second aim of this study is to evaluate usability and user adherence of the online/digital intervention through the Gokhale Method Foundation Class (online delivery with smartphone App).

The investigator hopes to learn:

The effectiveness of the Gokhale Method posture therapy for low back pain management, in comparison to the effectiveness of standard physical therapy with posture training.

the usability and user adherence of the online/digital intervention through the Gokhale Method Foundation Class (online delivery with smartphone App).

DETAILED DESCRIPTION:
100 participants with chronic low back pain will be recruited through the Stanford PMR clinics (Redwood City, Emeryville, Los Gatos, and Palo Alto). Information about the study will also be disseminated to the Stanford Primary Care clinics and through community advertisements.

Patients will be referred to the reaserch team by the providers who is been recommended for Physical Therapy.

Research team personnel will approach the recommended patients via email and will screen them prior to consenting for eligibility criteria by sending out a set of questionnaires via Redcap.

Eligible patients will be consented remotely via Redcap and will be subjected to randomization.

Eligible and consented participants will be randomly assigned (1:1) into one of the two intervention groups. Prior to intervention, participants will be asked to complete questionnaires on demographics, self-reported levels of pain, functional status, and disability levels. The questionnaires include:

Roland Morris Disability Questionnaire (RMDQ), Numeric Pain Rating Scale (NPRS), Patient-Reported Outcomes Measurement Information System (PROMIS-29),

Participants will be randomized (1:1) into the Gokhale method posture treatment (Gokhale) arm will receive a 18-sessions coaching under the Gokhale Elements course (may spread between 6-12 weeks, 1- 2 times per week, online delivery). Participants randomized into the standard care/physical therapy (PT) arm will similarly receive a standardized PT prescription during a 6-12 weeks period, meeting 1-2 times per week, to include posture education and training, therapeutic exercise instructions and development of an independent home exercise program.

Participants enrolled in the Gokhale Arm will be provided the Gokhale PostureTracker, a wearable posture monitoring sensor developed for interactive posture coaching, and a loaner smartphone with pre-installed App. Participants will be provided instruction to apply the sensor on their lumbar area and receive real-time visual feedback on their posture kinematic during the class. Participants can also perform normal daily activities while wearing the device. Data collected by the sensor will be sent to a HIPAA compliance server and shared with Stanford researchers.

Participant will complete remote follow-up assessments upon completion of their respective intervention, and at 6, and 12-month post intervention.

Primary outcomes assessed at baseline and each follow-up include the RMDQ,NPRS, PROMIS-29, PCS Secondary outcomes at each timepoint include 1) patient satisfaction and adherence. 2) Type, incidence and severity of complications and adverse events. 3) Concurrent pain medication use (including opioids) All collected data will be stored in a Stanford-secured server. No data would be transmitted to a third party. Access to the data will be limited exclusively to members of the research team.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old (working age population).
* NPRS score 4 or more for lower back.
* RMDQ score 7 and above.
* English speaking population
* Need insurance

Exclusion Criteria:

* Pregnancy (as stated by patient)
* With cognitive or communication impairment .
* Patients recommended for surgery
* Participating in other form of intervention.
* Prior history of chronic neurological disorder that impacts mobility (e.g. stroke, Parkinson's disease, multiple sclerosis)
* Fibromyalgia
* Underwent PT treatment for low back pain in the last 6 months
* Underlying mental disorder/untreated depression or presence of neurologic disorders such as MS, Alzheimers, Parkinsons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming in PM&R clinic with chronic lower back pain
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
NPRs ( national pain score) | 6-12 weeks
  Average pain score related to lower back
PROMIS-29 questionnaire | 6-12 weeks
  Patient-Reported Outcomes Measurement Information System
RMDQ questionnaire | 6-12 weeks
  Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
patient satisfaction and adherence | 12 months
  Post study evaluation of patient's satisfaction.
Type, incidence and severity of complications and adverse events | 12 months
Concurrent pain medication use (including opioids) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smuck, MD, Principal Investigator — Stanford PM&R Orthopedic surgery
Locations (1):
- Outpatient Surgery Center/Stanford Spine Clinic, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
Full data access will be limited to members of the research team.